CLINICAL TRIAL: NCT06001411
Title: Effect of Preoperative Prone Position Training on Postoperative Pulmonary Complications in Patients Undergoing Laparoscopic Colorectal Surgery
Brief Title: Effect of Prone Position Training on Pulmonary Complications in Patients Undergoing Laparoscopic Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Min Su (Other)
Responsible Party: Sponsor-Investigator, Min Su, Professor of Anesthesiology, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CQMUAZD2023
Record Dates: First submitted 2023-08-06; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Complication
Keywords: pulmonary complications, prone position , colorectal surgery
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Position Training group (PPT group) (Experimental): All patients were admitted to our hospital at least 3 days before surgery. Patients in the intervention group (PPT group) received the prone position training daily in the hospital, three times a day, and about 1 hours every times, for at least 3 days before surgery. On the day of admission to the hospital, the patients in the PPT group were instructed to perform prone position training by nurses who were previously trained by prone position training.
  Interventions: Behavioral: Prone Position Training
- Control group (C group) (Placebo Comparator): Patients in the control group (C group) received standard perioperative care without any prone position training.
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: Prone Position Training — All patients were admitted to our hospital at least 3 days before surgery. Patients in the intervention group (PPT group) received the prone position training daily in the hospital, three times a day, and about 1 hours every times, for at least 3 days before surgery. On the day of admission to the hospital, the patients in the PPT group were instructed to perform prone position training by nurses who were previously trained by prone position training.
  Arms: Prone Position Training group (PPT group)
Behavioral: control group — Patients in the control group (C group) received standard perioperative care without any prone position training.
  Arms: Control group (C group)

SUMMARY:
Colorectal cancer is a common digestive tract tumor in China. At present, laparoscopic surgery has become the classic operation of colorectal cancer surgery compared with the traditional open abdominal surgery. Although laparoscopic surgery has many advantages, such as less pain, faster recovery and so on. However, relevant studies have shown that postoperative pulmonary complications are more common in patients undergoing Laparoscopic Colorectal Surgery, which contribute to significant increases in morbidity, mortality, length of postoperative hospital stay and medical consumption.

The incidence of pulmonary complications after abdominal surgery has been reported to be between 9% and 40%.

The reduction in pulmonary volume and respiratory muscular activation after major abdominal surgery due to surgery-related shallow breathing, pain, long-term bed rest, mucociliary clearance disorder, and diaphragmatic dysfunction may be the main causes of postoperative pulmonary complications.

Numerous studies have demonstrated physiological improvement related to prone positioning. Prone positioning consists of placing a patient face down. Prone positioning has been used for to improve oxygenation in patients who require invasive mechanical ventilation for acute respiratory distress syndrome (ARDS). It has also been applied to non-intubated patients with acute respiratory failure (ARF), to improve oxygenation and delay or even avoid the need for invasive ventilation. So, the purpose of this study is to observe whether preoperative prone position training can reduce the incidence of pulmonary complications after laparoscopic colorectal cancer surgery.

DETAILED DESCRIPTION:
Colorectal cancer is a common digestive tract tumor in China. At present, laparoscopic surgery has become the classic operation of colorectal cancer surgery compared with the traditional open abdominal surgery. Although laparoscopic surgery has many advantages, such as less pain, faster recovery. However, relevant studies have shown that postoperative pulmonary complications are more common in patients undergoing Laparoscopic Colorectal Surgery, which contribute to significant increases in morbidity, mortality, length of postoperative hospital stay and medical consumption.

Postoperative pulmonary complications (PPCs) refer to the clinical abnormal changes in the lungs after surgery, These include lung infections (pneumonia), atelectasis, pleural effusion, bronchospasm, acute respiratory failure or acute respiratory distress syndrome (ARDS). The incidence of pulmonary complications after abdominal surgery has been reported to be between 9% and 40%.

The reduction in pulmonary volume and respiratory muscular activation after major abdominal surgery due to surgery-related shallow breathing, pain, long-term bed rest, mucociliary clearance disorder, and diaphragmatic dysfunction may be the main causes of postoperative pulmonary complications.

Numerous studies have demonstrated physiological improvement related to prone positioning. Prone positioning consists of placing a patient face down. Prone positioning has been used for more than 40 years to improve oxygenation in patients who require invasive mechanical ventilation for acute respiratory distress syndrome (ARDS). Because of the positive physiological effects of prone positioning on transpulmonary pressure, lung compression and ventilation perfusion ratio, it has also been applied to non-intubated patients with acute respiratory failure (ARF), to improve oxygenation and delay or even avoid the need for invasive ventilation.

Currently, the mechanisms of prone position training are decreased lung compression in the gravity dependant zone,homogenisation of transpulmonary pressure, improvement of ventilation/perfusion ratio, and reduction of ventilator-induced lung injury (VILI) or patient self-inflicted lung injury (P-SILI). By placing the patient in the prone position, the lungs compression due to its own weight is reduced via a gravitational-dependent redistribution of fluids. In addition, the weight of the mediastinum is supported by the sternum, the stiffer part of the chest. At the same time, the diaphragm is displaced caudally, decreasing compression of the posterior-caudal lung parenchyma. Finally, in a triangular-shaped lung, more parenchyma is included in the dorsal half than in the ventral one resulting in a more aerated lung in prone positioning.

So, the purpose of this study is to observe whether preoperative prone position training can reduce the incidence of pulmonary complications after laparoscopic colorectal cancer surgery.

This study was approved by the institutional review board of the First Affiliated Hospital of Chongqing Medical University. The protocol design is in accordance with Consolidated Standards of Reporting Trials (CONSORT) statement. All potentially eligible participants will be asked to give written informed consent before they are enrolled in this study. This study is a prospective, randomized, controlled clinical trial guided by the standard of good clinical practice (GCP), and eligible participants are divided into two groups: group PPT and group C, and primary assess the incidence of pulmonary complications after laparoscopic colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* Clinical diagnosis of colorectal cancer

Exclusion Criteria:

* Emergency surgery
* Cognitive dysfunction
* American Society of Anesthesiologists class ⩾IV
* Fractures (face, collarbone, ribs, spine, limbs)
* History of spontaneous pneumothorax
* Increased intracranial pressure
* pregnancy
* Systemic infection
* Acute respiratory failure
* Patients with hemodynamic instability
* Other conditions that are not suitable for prone position
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-08-21 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative pulmonary complications（PPCs） | 7 day after surgery
  The PPCs included pneumonia, atelectasis, pleural effusion, respiratory failure, and unplanned intubations

SECONDARY OUTCOMES:
arterial partial pressure of oxygen (PaO2) | preoperatively prior to starting prone position training, entering the operating room, the first day after surgery, the second day after surgery, and the third day after surgery
  Based on the blood gas analysis
extubation time | Day of surgery
  extubation time in postanesthesia care unit （PACU）
Peak airway pressure | Intraoperative
  Airway pressure
arterial partial pressure of carbon dioxide (PaCO2) | preoperatively prior to starting prone position training, entering the operating room, the first day after surgery, the second day after surgery, and the third day after surgery
  Based on the blood gas analysis
oxygenation index (OI) | preoperatively prior to starting prone position training, entering the operating room, the first day after surgery, the second day after surgery, and the third day after surgery
  Based on the blood gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, MD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- China,Chongqing The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China